CLINICAL TRIAL: NCT03365284
Title: Smart Kneebrace for Continuous Monitoring of Joint Angles During Rehabilitation After Total Knee Arthroplasty
Brief Title: Smart Kneebrace for Continuous Monitoring of Joint Angles During Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University (Other)
Responsible Party: Principal Investigator, Yifan Chen, Clinical professor ofarthritis clinic and research center, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUPHACRCE
Record Dates: First submitted 2017-11-25; First posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Arthroplasty, Replacement, Knee; Knee Osteoarthritis
Keywords: total knee arthroplasty; rehabilitation; Smart Kneebrace
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smart Kneebrace (Experimental): Smart Kneebrace with a smart phone app will be used during the rehabilitation after surgery for three months
  Interventions: Device: Smart Kneebrace with a smart phone app
- without Smart Kneebrace (Placebo Comparator): regular rehabilitation procedure will be applied after surgery
  Interventions: Other: regular rehabilitation procedure

INTERVENTIONS:
Device: Smart Kneebrace with a smart phone app — Smart Kneebrace will be used during the rehabilitation. Patients wearing the Smart KneeBrace are able to know their daily activity summary and exercise performance during rehabilitation training through a smart phone app.
  Arms: Smart Kneebrace
Other: regular rehabilitation procedure — regular rehabilitation procedure, especially muscle strengthening exercises
  Arms: without Smart Kneebrace

SUMMARY:
This study aims to investigate the effect of Smart Kneebrace use for osteoarthritis patients after total knee arhtroplasty (TKA) on post-operative performance.

DETAILED DESCRIPTION:
This is a single-center, open-label randomized controlled clinical trail. A total of 60 participants will receive total knee arthroplasty, who will be randomly assigned into experiment or control group. Smart Kneebrace will be used for the patients during the rehabilitation for the patients in experiment group, while the patients in the control group will not receive such a smart kneebrace. Postoperative joint angles as well as visual analog scale pain score, the Western Ontario and McMaster Universities Osteoarthritis Index knee society score will be estimated before operation and at 6/12 weeks after operation.

ELIGIBILITY:
Inclusion Criteria:

* Ready to receive single-side TKA

Exclusion Criteria:

* contraindication of surgery
* self-reported diseases that cause lower limb disability (for example, cerebrovascular disease especially stroke)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of postoperative joint angles | before operation and 6/12 weeks after operation
  Patients in both groups will wear the smart kneebrace by which the range of motion of the knee joint can be calculated.

SECONDARY OUTCOMES:
The change of knee pain. | before operation and 6/12 weeks after operation
  Visual Analogue Scale of pain is a scale to extimate pain, and its score ranges from 0 to 10. The higher the score is, the more severe pain the patient is feeling.
The change of knee symptoms. | before operation and 6/12 weeks after operation
  The Western Ontario and McMaster Universities Osteoarthritis Index(WOMAC),and its score ranges from 0 to 96. The higher the score is, the more severe symptoms the patient is feeling.

CONTACTS AND LOCATIONS:
Overall Officials: Jianhao Lin, MD, Principal Investigator — Arthritis clinic and research center, Peking University Peoples' Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel S, Park H, Bonato P, Chan L, Rodgers M. A review of wearable sensors and systems with application in rehabilitation. J Neuroeng Rehabil. 2012 Apr 20;9:21. doi: 10.1186/1743-0003-9-21. PMID 22520559
- [Background] Sosdian L, Dobson F, Wrigley TV, Paterson K, Bennell K, Dowsey M, Choong P, Allison K, Hinman RS. Longitudinal changes in knee kinematics and moments following knee arthroplasty: a systematic review. Knee. 2014 Dec;21(6):994-1008. doi: 10.1016/j.knee.2014.09.009. Epub 2014 Oct 12. PMID 25311517
- [Background] Mills K, Hunt MA, Ferber R. Biomechanical deviations during level walking associated with knee osteoarthritis: a systematic review and meta-analysis. Arthritis Care Res (Hoboken). 2013 Oct;65(10):1643-65. doi: 10.1002/acr.22015. PMID 23554153
- [Background] Brostrom EW, Esbjornsson AC, von Heideken J, Iversen MD. Gait deviations in individuals with inflammatory joint diseases and osteoarthritis and the usage of three-dimensional gait analysis. Best Pract Res Clin Rheumatol. 2012 Jun;26(3):409-22. doi: 10.1016/j.berh.2012.05.007. PMID 22867935